CLINICAL TRIAL: NCT05759741
Title: Alterations of Gut Microbiome, Function, and Its Intervention After Total Mesorectal Excision With Defunctioning Ileostomy for Mid-low Rectal Cancer
Brief Title: Alterations of Gut Microbiome, Function, and Its Intervention After Defunctioning Ileostomy
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Jianbin Xiang, Clinical Professor, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY2022-1095
Record Dates: First submitted 2023-02-12; First posted 2023-03-08 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Ileostomy - Stoma; Rectal Cancer; Microbial Disease; Intestinal Functional Disorder
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Intervention Model Description: The intervention group was given probiotics: 4 tablets of MIYAIRI 588, inserted into the distal ileostomy, once a week. The control group was not given drugs, only monthly outpatient follow-up of the anastomosis stoma.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MIYAIRI 588 group (Experimental): 4 tablets of MIYAIRI 588 were inserted into distal ileostomy once a week for 6 months.
  Interventions: Drug: MIYAIRI 588
- control group (No Intervention): The anastomosis stoma was followed up monthly in the outpatient department

INTERVENTIONS:
Drug: MIYAIRI 588 — 4 tablets of MIYAIRI 588 were inserted into the distal ileostomy once a week for 6 months
  Arms: MIYAIRI 588 group

SUMMARY:
This study focused on the alterations of gut microbiome and function during defunctioning ileostomy, and observed the effects of probiotic intervention on intestinal microbiome and function. The investigators looked forward to find the specific intestinal maladjusted flora from this work, which could provide a new scheme for the subsequent treatment of the damaged intestinal function and the reduction of the incidence of postoperative complication.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with primary rectal cancer received total mesolectal resection combined with defunctioning ileostomy.
2. Patients voluntarily sign informed consent.

Exclusion Criteria:

1. Disease progression or death after surgery.
2. Patients with inflammatory bowl disease.
3. Patients need to be on antibiotics/other probiotics for a long time.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2023-01-17 (Actual); Primary Completion 2024-07-17 (Estimated); Study Completion 2024-07-17 (Estimated)

PRIMARY OUTCOMES:
Wexner incontinence score | 1 year
  Assess defecation function，the score range is 0-20, 0 is normal, 20 is complete incontinence

SECONDARY OUTCOMES:
fecal incontinence quality-of-life scale | 1 year
  The Fecal Incontinence Quality of Life Scale is composed of a total of 29 items; these items form four scales: Lifestyle (10 items), Coping/Behavior (9 items), Depression/Self-Perception (7 items), and Embarrassment (3 items). The score of each scale is 1-4 points. The higher the score, the worse the quality of life.
Rate of postoperative complications | 1 month after operation
  Such as anastomotic leakage, operative death, intestinal obstruction, intestinal infection，etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan hospital, Shanghai, China